CLINICAL TRIAL: NCT06814301
Title: Impact of CMV-Specific Immune Reconstitution at the End of Letermovir Prophylaxis on the Development of Late Cytomegalovirus Infection in HSCT Recipients (INMUNOEND): a Protocol for a Prospective, Observational, Multicenter Study
Brief Title: Impact of CMV-Specific Immune Reconstitution at the End of Letermovir Prophylaxis on the Development of Late Cytomegalovirus Infection in Hematopoietic Stem Cell Transplant Recipients (INMUNOEND)
Acronym: INMUNOEND
Status: Not yet recruiting | Type: Observational
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Other Study IDs: FCO-INM-2024-04
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cytomegalovirus Cell Mediated Immunity; Stem Cell Transplantation, Hematopoietic
Keywords: stem cell transplantation; cytomegalovirus; letermovir; prophylaxis; cytomegalovirus immunity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 200 Days
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing allogenic-SCT who receive LTV prophylaxis with letermovir
  Interventions: Diagnostic Test: Periodic immunological monitoring of CMV-specific immune reconstitution will be performed using QTF-CMV

INTERVENTIONS:
Diagnostic Test: Periodic immunological monitoring of CMV-specific immune reconstitution will be performed using QTF-CMV — A first determination will be made pre-HCT, followed by subsequent determinations at +30, +60, +90, +120, +150, +180, and +200 days post-HCT, as well as at the end of prophylaxis with Letermovir
Diagnostic Test: Periodic immunological monitoring of CMV-specific immune reconstitution will be performed using QTF-CMV — A first determination will be made pre-HCT, followed by subsequent determinations at +30, +60, +90, +120, +150, +180, and +200 days post-HCT, as well as at the end of prophylaxis with LTV

SUMMARY:
Cytomegalovirus (CMV) infection is a common complication in patients undergoing hematopoietic stem cell transplantation (SCT). Fixed-duration letermovir (LTV) prophylaxis during the first 100 days post-SCT is effective and safe in preventing this infection, although it may be associated with a delay in CMV-specific immune reconstitution. Hence, it is needed a study to evaluate whether the absence of CMV-specific immune reconstitution at the end of LTV prophylaxis is associated with the development of late infection. This could facilitate the individualization of CMV prophylaxis duration in these patients.

Methods and analysis: INMUNOEND is a multicenter, prospective, observational, non-interventional study including CMV seropositive patients undergoing allo-SCT who receive LTV prophylaxis during the first 100 days post-SCT. Immunological and virological monitorization will be conducted until day +200 post-SCT. The primary outcome variable is the percentage of patients who develop clinically significant CMV infection up to day +200 post-SCT after completing LTV prophylaxis. Data collected will include: baseline characteristics of the hematological diseases and comorbidities, variables related to SCT (i.e. engrafment, graft-versus-host disease, use of letermovir and CMV replication) and variables related to CMV-specific immune reconstitution.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* CMV seropositivity (positive IgG) in the recipient at the time of SCT.
* First allogeneic hematopoietic stem cell transplant recipient (bone marrow, peripheral blood, or cord blood).
* Within the first 28 days post-SCT at the time of inclusion.
* Indication for LTV prophylaxis within the first 28 days post-transplant up to 100 days post-SCT, according to the criteria established in each center.

Exclusion Criteria:

* CMV seronegativity (negative IgG) in the recipient at the time of transplant.
* Previous allogeneic stem cell transplant (patients with a prior autologous transplant are allowed to be included).
* History of CMV disease in the 6 months prior to inclusion.
* Need for preemptive therapy in the month prior to inclusion in the study.
* Received any of the following in the 14 days prior to inclusion: Ganciclovir, valganciclovir, foscarnet, acyclovir (at doses >3200 mg orally per day or >25 mg/kg IV per day), valacyclovir (at doses >3000 mg orally per day), famciclovir (at doses >1500 mg orally per day).
* Received any of the following in the 30 days prior to screening: Cidofovir, CMV hyperimmune immunoglobulin, any CMV antiviral in the investigational phase.
* Suspected or confirmed hypersensitivity reaction to the LTV formulation or any of its components.
* Severe hepatic insufficiency (defined as Child-Pugh class C).
* History of primary immunodeficiency prior to transplant.
* Participation in a clinical trial involving the administration of CMV vaccines, other investigational CMV drugs, or monoclonal antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive CMV seropositive patients undergoing allogenic-SCT who receive LTV prophylaxis will be included. These patients will be prospectively evaluated during the first 200 days post-SCT.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
percentage of patients who develop clinically significant CMV infection (CMV-Cs) up to day +200 post-SCT after completing LTV prophylaxis | From enrollment to 200 days post-SCT

SECONDARY OUTCOMES:
proportion of patients with CMV-specific immune reconstitution at each QTF-CMV measurement point | From enrollment to 200 days post-SCT
proportion of patients with CMV replication during the 30 days following QTF-CMV testing | From enrollment to 200 days post-SCT
detection of any CMV replication and maximum copy number (IU/mL) during follow-up | From enrollment to 200 days post-SCT
percentage of patients without CMV-specific immune reconstitution at the end of LTV prophylaxis | From enrollment to 200 days post-SCT

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available after the end of the study
Supporting Information: Study Protocol, ICF
Time Frame: After publishing the results in a journal.
Access Criteria: Upon request to uicec@imibic.org

REFERENCES:
- [Derived] Caston JJ, Aparicio C, Paez-Vega A, Pozo Lopez L, Garcia E, Martin C, Ruiz-Arabi E, Cuesta-Casas MA, Bermudez-Rodriguez MA, Cerezo-Martin JM, Gonzalez-Sierra PA, Machuca I, Martin Dominguez FM, Saldana-Moreno R, Herrera C, Torre-Cisneros J. Impact of CMV-specific immune reconstitution at the end of letermovir prophylaxis on the development of late cytomegalovirus infection in haematopoietic stem cell transplant recipients (INMUNOEND): a protocol for a prospective, observational, multicentre study. BMJ Open. 2025 Oct 15;15(10):e101289. doi: 10.1136/bmjopen-2025-101289. PMID 41093321